CLINICAL TRIAL: NCT06328517
Title: The Influence of Nutritional Factors on the Prognosis of Liver Cirrhosis Patients and the Exploration of Predictive Models
Status: Recruiting | Type: Observational
Sponsor: Juan Kang (Other)
Responsible Party: Sponsor-Investigator, Juan Kang, associate professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2023-305
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cirrhosis
Keywords: rest energy expenditure; malnutrition; prognosis
MeSH Terms: conditions — Fibrosis; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with cirrhosis: Abdominal ultrasound, CT, or MRI showed Cirrhosis during the screening period; Fibroscan results during the screening period were> 17.5kPa.

SUMMARY:
Cirrhosis is a progressive developing liver disease transforming normal hepatocytes into scar tissue with loss of function.The prevalence of cirrhosis has approximately tripled over the past two decades. With the increasing incidence of chronic liver disease, about 2 million people died from cirrhosis worldwide. Currently, D'Amico stage classification and Child-Pugh and Model for End-Stage Liver Disease (MELD) scores constitute the best tools to predict mortality in patients with Cirrhosis; however, one of their main limitations is the lack of evaluation of the nutritional and functional status. Patients with End-Stage Liver Disease (ESLD) have reduced nutritional intake, hypermetabolism, increased energy expenditure, impaired fasting adaptability, decreased hepatic glycogen reserves, and increased consumption of protein as the main energy donor that often lead to malnutrition, therefore, malnutrition is one of the most common complications in patients with Cirrhosis, is closely related to the increase in morbidity and mortality. Moreover, malnutrition is closely related to the high incidence of infection, ascites, hepatic encephalopathy, and hepatorenal syndrome, and is an independent risk factor affecting the survival rate of patients with End-Stage Liver Disease, including liver transplantation.

Therefore, malnutrition should be treated as equally important complications such as ascites and hepatic encephalopathy, and accurate screening, evaluation and appropriate nutritional intervention measures should be taken to improve the prognosis of patients with Cirrhosis. This study aims to establish a nomogram model about nutritional factors to predict the prognosis of patients with Cirrhosis, verify and optimize the model, through the establishment of the model, to more comprehensively evaluate and predict the prognosis of patients with Cirrhosis from the perspective of nutrition, to provide sufficient basis and lay a solid foundation for further nutritional intervention and improve patient prognosis.

DETAILED DESCRIPTION:
Patients with Cirrhosis attending the Second Affiliated Hospital of Chongqing Medical University were included in the retrospective study. Participants met the inclusion and exclusion criteria. The data to be collected include basic information including gender, age, height and weight; blood routine, liver and kidney function, coagulation function, abdominal CT / MRI, underlying disease, complications, treatment options, disease changes, etc; professional Resting Energy Expenditure (REE) measurement and regular follow-up. After the data collection, the effects of REE, albumin, 2,5-OH vitamin D, and muscle function on the long-term prognosis of the patients with Cirrhosis were investigated by drawing the survival curve, the Receiver-Operating Characteristic curve (ROC curve) , and the Area Under a ROC curve (AUC curve) .

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign an informed consent form;
2. Abdominal ultrasound, CT, or MRI showed cirrhosis during the screening period; Fibroscan results during the screening period were> 17.5kPa;
3. Estimated survival time of more than 3 months;
4. Full capacity for civil conduct.

Exclusion Criteria:

1. The diagnosis of primary liver cancer or was supported by the following evidence: increased alpha-fetoprotein (AFP) (≥100 μg/L) for more than 3 months or liver imaging showed clear liver cancer nodules in the liver;
2. A history of malignancy within 5 years prior to screening, except for specific cancers (such as basal cell skin cancer); current or prior history of major disease that may interfere with personal treatment, assessment or compliance. Major diseases are 25 major diseases as stipulated by the China Insurance Regulatory Commission;
3. Severe lung disease, severe heart disease, diabetes mellitus, or genetic and metabolic diseases;
4. Psychiatric hospitalization, attempted suicide, and / or temporary disability due to mental illness in the past five years;
5. Pregnant or lactating women;
6. The investigator considered not unsuitable for participants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Abdominal ultrasound, CT, or MRI showed cirrhosis during the screening period; Fibroscan results during the screening period were> 17.5kPa.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Death | January 2024 to November 2026
  Death due to cirrhosis progression

SECONDARY OUTCOMES:
complication | January 2024 to November 2026
  complication such as infection, ascites.

CONTACTS AND LOCATIONS:
Overall Officials: juan Kang, M.D., Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China